CLINICAL TRIAL: NCT05035927
Title: A Phase 2a Safety and Feasibility Study Evaluating Psilocybin (TRP-8802) Administration in Concert With Psychotherapy in the Treatment of Binge Eating Disorder
Brief Title: Evaluation of Psilocybin (TRP-8802) in the Treatment of Binge Eating Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TRYP Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRYP-001
Record Dates: First submitted 2021-08-24; First posted 2021-09-05 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Binge Eating Disorder
MeSH Terms: conditions — Binge-Eating Disorder | interventions — Psilocybin; Psychotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open Label Oral Psilocybin (Experimental)
  Interventions: Drug: TRYP-0082; Behavioral: Psychotherapy

INTERVENTIONS:
Drug: TRYP-0082 — A single (1) 25 mg oral dose of TRP 8802 will be administered in a carefully monitored setting following 6 to 8 hours of preparatory psychotherapy. Subjects will be in the study for 12 weeks following the dose of TRP 8802 (until Week 14), approximately 5 months from initiation of screening through the last follow-up.
  Other Names: Psilocybin
Behavioral: Psychotherapy — A single (1) 25 mg oral dose of TRP 8802 will be administered in a carefully monitored setting following 6 to 8 hours of preparatory psychotherapy. Subjects will be in the study for 12 weeks following the dose of TRP 8802 (until Week 14), approximately 5 months from initiation of screening through the last follow-up.

SUMMARY:
To better understand the potential benefits of psychedelics in overeating disorders, Tryp Therapeutics will conduct a safety and feasibility clinical trial using TRP 8802 among individuals with Binge Eating Disorder. This is a single-center phase 2a open-label study to assess the safety and feasibility of a single dose of TRP 8802 in subjects with BED. Subjects will undergo screening, preparation therapy sessions, dosing, integration therapy sessions, and follow-up for 12 weeks following the dose of TRP 8802. The total participation in the study will be up to approximately 5 months.

DETAILED DESCRIPTION:
Binge eating disorder is the most common eating disorder and is associated with obesity and psychiatric comorbidities, including depression, and impulsive and compulsive disorders. Binge eating disorder is marked by severe disturbance to a person's control over their eating behaviors and high anxiety around food. Various programs using psilocybin paired with psychotherapy have shown positive effects in treating a variety of psychiatric and behavioral conditions, including cancer-related psychiatric distress, anxiety, treatment-resistant depression, and nicotine and alcohol addiction. Based on clinical precedents, relevant neuropharmacology, and mechanistic similarities, psilocybin is theorized to have the potential to be part of the treatment of overeating disorders. TRP-8802 could accomplish this by moderating overall anxiety, anxiety around food, perseveration, and repetitive and intrusive thoughts about food in people with BED.

The primary objective of this study is to:

1. Assess the safety of a single dose of TRP 8802 in participants with binge eating disorder (BED) during the TRP 8802 dosing session, and through 12 weeks following dosing (i.e., Week 14).

ELIGIBILITY:
Inclusion/Exclusion Criteria: Inclusion Criteria:

To participate in this study, subjects will have to meet all of the following criteria:

1. Meet Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria for BED.
2. Age ≥18 and ≤64 years.
3. Provision of signed and dated informed consent form.
4. Stated willingness to comply with all study procedures and availability for the duration of the study.
5. Medically stable in the judgment of the Principal Investigator, as determined by screening medical, physical examination, ECG, and routine laboratory tests including blood and urinalysis.
6. For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation and for an additional 4 weeks following the dose of TRP 8802. Adequate birth control methods include intrauterine device; injected, implanted, intravaginal, or transdermal hormonal method; oral hormones plus a barrier contraception; abstinence; vasectomized sole partner; or double barrier contraception.
7. For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner through 90 days post-dose.
8. Agree to consume approximately the same amount of caffeine-containing beverage (e.g., coffee, tea) that he/she consumes on a usual morning, before arriving at the research unit on the morning of the drug session day. If the participant does not routinely consume caffeinated beverages, he/she must agree not to do so on the dosing session day.
9. Agree to refrain from using any psychoactive drugs, including alcoholic beverages for a minimum of 1 week prior to drug administration.
10. Agree that for 1 week before the drug session, including the morning of the session, he/she will refrain from taking any nonprescription medication, nutritional supplement, herbal supplement, or as needed (PRN) prescription medication except when approved by the study investigators. Exceptions will be evaluated by the study investigators and will include acetaminophen, non-steroidal anti-inflammatory drugs, and common doses of vitamins and minerals and contraceptives.

Exclusion Criteria:

To participate in this study, subjects must not meet any of the following criteria:

1. Significant suicide risk as defined by either suicidal ideation as endorsed on items 4 or 5 on the C-SSRS within the past year, at Screening, or at Baseline; or suicidal behaviors within the past year; clinical assessment of significant suicidal risk during subject interview.
2. Participation in another concurrent clinical study or within the preceding month.
3. Women who are pregnant or who intend to become pregnant during the study or who are currently nursing.
4. Vital signs, averaged over 3 readings within 15 minutes, of systolic blood pressure (BP) >139 mm Hg, diastolic BP >89 mm Hg, or heart rate >90 bpm.
5. Have any of the following cardiovascular conditions: uncontrolled hypertension, coronary artery disease, congenital long QT syndrome, cardiac hypertrophy, cardiac ischemia, congestive heart failure, prior myocardial infarction, tachycardia, artificial heart valve, QTc >450 msec at screening, any other clinically significant screening ECG abnormality, or any other significant cardiovascular condition.
6. Presence of a gastrointestinal disease that could interfere with absorption of orally-administered TRP 8802.
7. Have epilepsy.
8. Meet DSM-5 criteria for schizophrenia spectrum or other psychotic disorders, including major depressive disorder with psychotic features, or Bipolar I or Bipolar II Disorder.
9. Family history of psychosis.
10. Meet DSM-5 criteria for a moderate or severe alcohol or drug use disorder.
11. Positive urine drug screen or alcohol breath test at screening. A repeat test can be conducted at screening or Day -1 at the discretion of the Principal Investigator or delegate.
12. Prior adverse effects from psilocybin.
13. Currently taking or expected to need prior to the dosing session, UGT1A9 or 1A10 inhibitors (e.g., regorafenib, rifampicin, phenytoin, eltrombopag, mefenamic acid, diflunisal, niflumic acid, sorafenib, isavuconazole, deferasirox, ginseng) and aldehyde or alcohol dehydrogenase inhibitor (e.g., disulfiram).
14. Currently taking or testing positive on urine drug screen, drugs of abuse such as amphetamines, buprenorphine, benzodiazepines, cocaine, methamphetamines, Ecstasy (MDMA), morphine, methadone, oxycodone, marijuana, ethyl glucuronide, fentanyl, tramadol, and synthetic cannabinoids (K2).
15. Currently taking on a regular (e.g., daily) basis any medications having a primary centrally-acting serotonergic effect, including SSRIs, MAOIs, or serotonin-acting dietary supplements (such as 5 hydroxy tryptophan or St. John's wort). For individuals who have intermittent or PRN use of such medications, the dosing session will not be conducted until at least 5 half-lives of the agent have elapsed after the last dose.
16. fMRI subjects: Contraindications to fMRI procedures, per institutional policy.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2024-03-07 (Actual); Study Completion 2024-06-07 (Actual)

PRIMARY OUTCOMES:
Assess the safety of a single dose of TRP 8802 in participants with BED during the TRP 8802 dosing session, and through 12 weeks following dosing | 12 weeks following dosing
  Safety assessments will be conducted to monitor AEs, including SAEs, protocol specific safety laboratory assessments, protocol specific vital signs and other tests/questionnaires that are deemed crucial to the safety evaluation of the study. Planned timing for all safety assessments is provided in the SOA.

SECONDARY OUTCOMES:
Evaluate the feasibility of inducing the psychedelic state with TRP 8802 in a BED population. | 12 weeks following dosing
  Magnitude and duration of TRP 8802-induced dissociative effects in participants with BED using the MEQ30 and MRS
Determine the preliminary clinical activity and the effects of TRP 8802 in conjunction with psychotherapy on the frequency of binge eating episodes in a BED population through 4 weeks following dosing (i.e., Week 6) | 6 Weeks
  Frequency of binge eating episodes as measured by a modified Eating Questionnaire
Determine the preliminary clinical activity and the effects of TRP 8802 in conjunction with psychotherapy on weight-related indicators in a BED population through 4 weeks following dosing (i.e., Week 6) | 6 Weeks
  Waist Circumference and BMI

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Miller, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No